CLINICAL TRIAL: NCT04808531
Title: NanaBis™ an Oro-buccal Administered Equimolar d9-THC & CBD Formulation as Monotherapy for Management of Opioid Requiring Bone Pain Due to Metastatic Cancer: Phase 3 Multi Centre Blinded Randomized Withdrawal Active & Placebo Controlled Trial
Brief Title: NanaBis™ an Oro-buccal Administered delta9-Tetrahydrocannabinol (d9-THC) & Cannabidiol (CBD) Medicine for the Management of Bone Pain From Metastatic Cancers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medlab Clinical (Industry)
Collaborators: Emerald Clinical Inc. (Industry); WriteSource Medical Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDC-NB-P3-01
Record Dates: First submitted 2021-03-11; First posted 2021-03-22 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Cancer Related Pain
Keywords: Cannabis based medicine; d9-tetrahydrocannabinol; Cannabidiol; Cancer Pain; Cancer Bone Pain; Treatment; Monotherapy; Nanoparticle; Tetrahydrocannabinol
MeSH Terms: conditions — Cancer Pain | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple blinding
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double Placebo Arm (Placebo Comparator): Spray Placebo + Tablet Placebo
  Spray Placebo is a nanoparticle water soluble solution without cannabinoids containing a small amount of hemp seed oil (for fragrance purposes only) as defined by Australian Office of Drug Control (ODC) (https://www.odc.gov.au/hemp-products). One dose is equivalent to 2 actuations of the pump delivering 280 µL volume.
  Tablet Placebo will be identical to the Oxycontin tablets.
  Interventions: Drug: Placebo Spray; Drug: Placebo Tablet; Drug: Oxycodone IR
- Treatment NanaBis™ Arm (Experimental): NanaBis™ + Tablet Placebo
  NanaBis™ is a nanoparticle water soluble equimolar solution of d9-THC and CBD. One dose is equivalent to 2 actuations of the pump delivering 280 µL volume containing 2.5 mg d9-THC and 2.5 mg CBD. The dose administered will be 1 - 3.5 doses (2 sprays to 7 sprays) per 4 hours unless asleep.
  Interventions: Drug: NanaBis™; Drug: Placebo Tablet; Drug: Oxycodone IR
- Comparator (Oxycodone) Arm (Active Comparator): Spray Placebo + Oxycodone CR
  Spray Placebo is a nanoparticle water soluble solution without cannabinoids containing a small amount of hemp seed oil (for fragrance purposes only) as defined by Australian ODC (https://www.odc.gov.au/hemp-products). One dose is equivalent to 2 actuations of the pump delivering 280 µL volume.
  Oxycodone controlled release (CR) used as a comparator will be Oxycontin tablets 10 mg - 70 mg po bd.
  Interventions: Drug: Oxycodone CR; Drug: Placebo Spray; Drug: Oxycodone IR

INTERVENTIONS:
Drug: NanaBis™ — NanaBis™ is a nanoparticle water soluble equimolar solution of d9-THC & CBD. One dose is equivalent to 2 actuations of the pump delivering 280 µL volume containing 2.5 mg d9-THC and 2.5 mg CBD
  Other Names: MDCNB-01; NanoCelle® d9-THC & CBD
  Arms: Treatment NanaBis™ Arm
Drug: Oxycodone CR — Oxycodone CR tablet is an opioid agonist supplied in 10 mg, 15 mg, 20 mg, 30 mg,40 mg, 60 mg and 80 mg tablets for oral administration. The tablet strengths describe the amount of oxycodone per tablet as the hydrochloride salt.
  Other Names: OxyNorm®; OxyContin®; Endone®; Proladone®; Targin®; Xtampza ER®
  Arms: Comparator (Oxycodone) Arm
Drug: Placebo Spray — Placebo comparator used against both NanaBis™ and Oxycodone depending on randomisation of arms.
  Other Names: NanoCelle® Placebo Spray
  Arms: Comparator (Oxycodone) Arm; Double Placebo Arm
Drug: Placebo Tablet — Placebo comparator used against both NanaBis™ and Oxycodone depending on randomisation of arms.
  Arms: Double Placebo Arm; Treatment NanaBis™ Arm
Drug: Oxycodone IR — Oxycodone immediate release (IR) tablet or capsule or oral solution used as breakthrough analgesia.
  Other Names: Oxyfast®; Oxy IR®; Oxaydo®; Roxicodone®

SUMMARY:
This is a multi-centre, long term, double blind, clinical protocol for NanaBis™ as a monotherapy treatment in participants 18-75 years of age with cancer related pain.

DETAILED DESCRIPTION:
This trial uses an alternative method to demonstrate the analgesic efficacy of NanaBis™ as a monotherapy in cancer participants. Proving analgesic efficacy requires demonstrating that (i) the analgesic is significantly better than placebo and (ii) that the magnitude of the improvement is clinically important. The latter is standardly done by measuring the change in pain levels from a baseline (no analgesia) to the end of a treatment period. A 30% decrease in the Numerical Pain Rating Scale (NPRS) has been correlated with participants reporting a moderate improvement in their pain and this was adopted as the standard method of demonstrating a clinically important magnitude of improvement. In this strategy, the measure of analgesic efficacy is the proportion of participants in the treatment group whose pain is adequately treated (responders). A responder is defined as a patient who completes the treatment phase with an acceptable level of pain (NPRS ≤ 5) and without requiring excessive amounts of rescue (breakthrough analgesia) medication. Unlimited breakthrough analgesia (Oxycodone) is allowed throughout the study; however, excessive use will result in discontinuation. Comparison of the proportion of responders in the NanaBis™ arm and placebo arms will determine if NanaBis™ is significantly better than placebo. Demonstrating that the proportion of responders in the NanaBis™ arm is non-inferior to the Oxycodone controlled release (CR) comparator arm will determine if the magnitude of improvement (provided by NanaBis™) is clinically important because Oxycodone CR has been established as the benchmark analgesic that provides a clinically important effect.

ELIGIBILITY:
Inclusion Criteria:

At Screening Phase

Participants must fulfil all of the following criteria:

* Prospective male and female participants that are:

  1. in the age range 18-65 years or
  2. 65 to 75 years without significant co-morbidities (heart, lung, liver or renal failure, myocardial infarction, cerebral vascular accident, peripheral vascular disease, chronic obstructive pulmonary disease, dementia, connective tissue disease or diabetes mellitus with end-organ damage)
* Metastatic bone pain from a cancer diagnosis is the only major cause of pain.
* Documented proof (imaging) confirming the Metastatic Bone Disease at the current site of pain and that there has no been treatment since diagnosis
* Meet International Classification of Diseases, Tenth Revision (ICD-10) codes for pain management criteria (i.e., bone cancer pain)
* During the screening period, the participant is on stable opioid pain management and pain severity (NPRS) ≤ 8 with a maximum variation of ± 1
* Pain Detect score > 18
* Participant willing and able to provide informed consent and follow study procedures

  1. including agreeing to not drive or operate heavy machinery; and
  2. females of child-bearing potential agree to use reliable contraception during the duration of the clinical trial
* Patient deemed tolerable to Oxycodone and NanaBis™ determined by medical history of allergies to cannabinoids or opioids
* Patient must not be a participant in a clinical trial or study.

Exclusion Criteria:

At Screening Phase

Participants will be excluded if they meet any of the following criteria that include:

* History of epilepsy or recurrent seizures
* Moderate to severe medical conditions such as

  1. Severe hepatic, cardiovascular, pulmonary or renal impairment or
  2. Psychiatric disorders (i.e., unstable schizophrenia, recent drug-induced psychosis, severe mood disorders), that would be assessed at the medical screen
* If participants have been diagnosed with a current substance abuse disorder
* Women who are pregnant, lactating or planning to become pregnant
* Identified concerns by the nursing / medical team relevant to the safe storage of medications (i.e., NanaBis™ or standard medical therapy)
* Participants who may not be available for follow up (i.e., planned or expected travel or other)
* Participants plan to undergo any treatment that will substantially reduce the burden of disease (and therefore bone pain) during the screening, titration or maintenance phase of the clinical trial such as radiotherapy or cytotoxic chemotherapy
* Participants who are unable to withhold all analgesia (apart from which is part of this trial) during the titration and maintenance phase of the study, including bisphosphonates, or are currently exceeding equivalence of 70mg BD Oxycodone CR. Medications such as bisphosphonates may be coordinated so they are given either side of the excluded period that covers the titration and maintenance phases
* Participants will NOT be excluded if they are being treated with maintenance pharmacotherapy to prevent progression of disease such as steroids and hormone therapy, which may be continued during the trial at a stable dose
* Participant will be excluded if they are participating in any other clinical trial or study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Significant changes in responders with NanaBis™ spray over placebo (p<0.05) | 6 weeks
  To demonstrate that at the end of the 6-week study period the proportion of responders in the NanaBis™ group shows significant change than the proportion of responders in the placebo group.
  A responder is defined as a participant who completes the maintenance phase with an acceptable level of pain (NPRS is equal to 5) and without requiring excessive amounts of rescue (breakthrough analgesia) medication.
  NPRS Assessment [Time Frame: Baseline and then twice daily for the duration of the study].
  The NPRS questionnaire is completed by the participant to determine their pain intensity. The NPRS is an 11-point scale scored from '0-10'. A score of '0' being no pain and a score of '10' being the most intense pain imaginable. Participants select the value that is most in line with the intensity of pain they have experienced in the last 24 hours.

SECONDARY OUTCOMES:
Comparable efficacy in proportion of responders from NanaBis™ spray to the proportion of responders to Oxycodone CR | 6 weeks
  To demonstrate that at the end of the 6-week study period the proportion of responders in the NanaBis™ group is similar to the proportion of responders in the Oxycodone group determined by pain levels recorded using NPRS.
  A responder is defined as a participant who completes the maintenance phase with an acceptable level of pain (NPRS is equal to 5) and without requiring excessive amounts of rescue (breakthrough analgesia) medication.
  NPRS Assessment [Time Frame: Baseline and then twice daily for the duration of the study].
  The NPRS questionnaire is completed by the participant to determine their pain intensity. The NPRS is an 11-point scale scored from '0-10'. A score of '0' being no pain and a score of '10' being the most intense pain imaginable. Participants select the value that is most in line with the intensity of pain they have experienced in the last 24 hours.
Significant change in the Health-Related Quality of Life Scores with NanaBis™ spray over placebo (p<0.05) and comparable to Oxycodone CR | 6 weeks
  To demonstrate that at the end of the 6-week study period the Health-Related Quality of Life scores in the NanaBis™ treated group are significantly changed than in the Placebo group and is similar to the Oxycodone CR treated group.
  Quality of life as assessed by the EORTC-QLQ-C30 validated questionnaire [ Time Frame: Baseline and then weekly during the maintenance phase of the study and at then weeks 7 and 18 of the Open Label Extension].
  The EORTC-QLQ-C30 is validated questionnaire answered by participants to assess the quality of life of cancer patients. It assesses important functioning domains (e.g. physical, emotional, role) and common cancer symptoms (e.g. fatigue, pain, nausea/vomiting, appetite loss).
Significant change in the NPRS score with NanaBis™ spray over placebo (p<0.05) and comparable to Oxycodone CR | 18 weeks
  NPRS Assessment [Time Frame: Baseline and then twice daily for the duration of the study].
  The NPRS questionnaire is completed by the participant to determine their pain intensity. The NPRS is an 11-point scale scored from '0-10'. A score of '0' being no pain and a score of '10' being the most intense pain imaginable. Participants select the value that is most in line with the intensity of pain they have experienced in the last 24 hours.
NanaBis™ Adverse Events | 18 weeks
  To demonstrate that at the end of the 6-week study period that NanaBis™ is safe and tolerable.
  Safety and tolerability will be assessed via standardised adverse events, Serious adverse events, Deaths, UKU - Side Effects Rating Scale (UKU), Local Adverse Events Charts and patient medical records.
  Adverse events, serious adverse events and deaths will be summarised by treatment arm.
  Does the daily use of NanaBis™ oro-buccal spray reduce the severity of Treatment-Emergent Adverse Events (safety and tolerability). [Time Frame: Baseline and then weekly for the duration of the study].
  Changes in validated UKU scale range is 0 to 3 for rating the degree of severity (mild, moderate or severe) and a second scale for the investigator that assigns a casual relationship of improbable, possible or probable.
Fifty percent or greater of the NanaBis™ treated group request compassionate extension with NanaBis™ spray | 12 weeks
  To demonstrate that at the end of the 6-week study period that after unblinding, half or more of the NanaBis™ treated group prefer further treatment with NanaBis™ in the open label extension phase (note that all participants will be all offered open label extension if appropriate).

REFERENCES:
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Kress HG, Koch ED, Kosturski H, Steup A, Karcher K, Lange B, Dogan C, Etropolski MS, Eerdekens M. Tapentadol prolonged release for managing moderate to severe, chronic malignant tumor-related pain. Pain Physician. 2014 Jul-Aug;17(4):329-43. PMID 25054392
- [Background] Anderson W. 2007 National Statement on Ethical Conduct in Human Research. Intern Med J. 2011 Jul;41(7):581-2. doi: 10.1111/j.1445-5994.2011.02528.x. No abstract available. PMID 21762341
- [Background] Portenoy RK. Treatment of cancer pain. Lancet. 2011 Jun 25;377(9784):2236-47. doi: 10.1016/S0140-6736(11)60236-5. PMID 21704873
- [Background] Deandrea S, Montanari M, Moja L, Apolone G. Prevalence of undertreatment in cancer pain. A review of published literature. Ann Oncol. 2008 Dec;19(12):1985-91. doi: 10.1093/annonc/mdn419. Epub 2008 Jul 15. PMID 18632721
- [Background] Wiffen PJ, McQuay HJ. Oral morphine for cancer pain. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD003868. doi: 10.1002/14651858.CD003868.pub2. PMID 17943804
- [Background] Kane CM, Hoskin P, Bennett MI. Cancer induced bone pain. BMJ. 2015 Jan 29;350:h315. doi: 10.1136/bmj.h315. No abstract available. PMID 25633978
- [Background] Gregorian RS Jr, Gasik A, Kwong WJ, Voeller S, Kavanagh S. Importance of side effects in opioid treatment: a trade-off analysis with patients and physicians. J Pain. 2010 Nov;11(11):1095-108. doi: 10.1016/j.jpain.2010.02.007. Epub 2010 May 10. PMID 20452835
- [Background] Macedo F, Ladeira K, Pinho F, Saraiva N, Bonito N, Pinto L, Goncalves F. Bone Metastases: An Overview. Oncol Rev. 2017 May 9;11(1):321. doi: 10.4081/oncol.2017.321. eCollection 2017 Mar 3. PMID 28584570
- [Background] Choong PF. The molecular basis of skeletal metastases. Clin Orthop Relat Res. 2003 Oct;(415 Suppl):S19-31. doi: 10.1097/01.blo.0000093839.72468.da. PMID 14600589
- [Background] Pezaro C, Omlin A, Lorente D, Rodrigues DN, Ferraldeschi R, Bianchini D, Mukherji D, Riisnaes R, Altavilla A, Crespo M, Tunariu N, de Bono J, Attard G. Visceral disease in castration-resistant prostate cancer. Eur Urol. 2014 Feb;65(2):270-273. doi: 10.1016/j.eururo.2013.10.055. Epub 2013 Nov 22. PMID 24295792
- [Background] Bubendorf L, Schopfer A, Wagner U, Sauter G, Moch H, Willi N, Gasser TC, Mihatsch MJ. Metastatic patterns of prostate cancer: an autopsy study of 1,589 patients. Hum Pathol. 2000 May;31(5):578-83. doi: 10.1053/hp.2000.6698. PMID 10836297
- [Background] Yanae M, Fujimoto S, Tane K, Tanioka M, Fujiwara K, Tsubaki M, Yamazoe Y, Morishima Y, Chiba Y, Takao S, Komoike Y, Tsurutani J, Nakagawa K, Nishida S. Increased risk of SSEs in bone-only metastatic breast cancer patients treated with zoledronic acid. J Bone Oncol. 2017 Aug 31;8:18-22. doi: 10.1016/j.jbo.2017.08.004. eCollection 2017 Sep. PMID 28884071
- [Background] Body JJ, Quinn G, Talbot S, Booth E, Demonty G, Taylor A, Amelio J. Systematic review and meta-analysis on the proportion of patients with breast cancer who develop bone metastases. Crit Rev Oncol Hematol. 2017 Jul;115:67-80. doi: 10.1016/j.critrevonc.2017.04.008. Epub 2017 Apr 23. PMID 28602171
- [Background] Coleman RE. Clinical features of metastatic bone disease and risk of skeletal morbidity. Clin Cancer Res. 2006 Oct 15;12(20 Pt 2):6243s-6249s. doi: 10.1158/1078-0432.CCR-06-0931. PMID 17062708
- [Background] Colloca L, Ludman T, Bouhassira D, Baron R, Dickenson AH, Yarnitsky D, Freeman R, Truini A, Attal N, Finnerup NB, Eccleston C, Kalso E, Bennett DL, Dworkin RH, Raja SN. Neuropathic pain. Nat Rev Dis Primers. 2017 Feb 16;3:17002. doi: 10.1038/nrdp.2017.2. PMID 28205574
- [Background] Murnion BP. Neuropathic pain: current definition and review of drug treatment. Aust Prescr. 2018 Jun;41(3):60-63. doi: 10.18773/austprescr.2018.022. Epub 2018 Jun 1. No abstract available. PMID 29921999
- [Background] Mantyh PW. Bone cancer pain: from mechanism to therapy. Curr Opin Support Palliat Care. 2014 Jun;8(2):83-90. doi: 10.1097/SPC.0000000000000048. PMID 24792411
- [Background] Ahmad I, Ahmed MM, Ahsraf MF, Naeem A, Tasleem A, Ahmed M, Farooqi MS. Pain Management in Metastatic Bone Disease: A Literature Review. Cureus. 2018 Sep 11;10(9):e3286. doi: 10.7759/cureus.3286. PMID 30443456
- [Background] Meng H, Johnston B, Englesakis M, Moulin DE, Bhatia A. Selective Cannabinoids for Chronic Neuropathic Pain: A Systematic Review and Meta-analysis. Anesth Analg. 2017 Nov;125(5):1638-1652. doi: 10.1213/ANE.0000000000002110. PMID 28537982
- [Background] Cavalli E, Mammana S, Nicoletti F, Bramanti P, Mazzon E. The neuropathic pain: An overview of the current treatment and future therapeutic approaches. Int J Immunopathol Pharmacol. 2019 Jan-Dec;33:2058738419838383. doi: 10.1177/2058738419838383. PMID 30900486
- [Background] Lee-Kubli CA, Calcutt NA. Painful neuropathy: Mechanisms. Handb Clin Neurol. 2014;126:533-57. doi: 10.1016/B978-0-444-53480-4.00034-5. PMID 25410243
- [Background] Deshpande A, Mailis-Gagnon A, Zoheiry N, Lakha SF. Efficacy and adverse effects of medical marijuana for chronic noncancer pain: Systematic review of randomized controlled trials. Can Fam Physician. 2015 Aug;61(8):e372-81. PMID 26505059
- [Background] Blake A, Wan BA, Malek L, DeAngelis C, Diaz P, Lao N, Chow E, O'Hearn S. A selective review of medical cannabis in cancer pain management. Ann Palliat Med. 2017 Dec;6(Suppl 2):S215-S222. doi: 10.21037/apm.2017.08.05. Epub 2017 Aug 23. PMID 28866904
- [Background] Ligresti A, De Petrocellis L, Di Marzo V. From Phytocannabinoids to Cannabinoid Receptors and Endocannabinoids: Pleiotropic Physiological and Pathological Roles Through Complex Pharmacology. Physiol Rev. 2016 Oct;96(4):1593-659. doi: 10.1152/physrev.00002.2016. PMID 27630175
- [Background] Sun J, Zhou YQ, Chen SP, Wang XM, Xu BY, Li DY, Tian YK, Ye DW. The endocannabinoid system: Novel targets for treating cancer induced bone pain. Biomed Pharmacother. 2019 Dec;120:109504. doi: 10.1016/j.biopha.2019.109504. Epub 2019 Oct 15. PMID 31627091
- [Background] Mao Y, Huang Y, Zhang Y, Wang C, Wu H, Tian X, Liu Y, Hou B, Liang Y, Rong H, Gu X, Ma Z. Cannabinoid receptor 2-selective agonist JWH015 attenuates bone cancer pain through the amelioration of impaired autophagy flux induced by inflammatory mediators in the spinal cord. Mol Med Rep. 2019 Dec;20(6):5100-5110. doi: 10.3892/mmr.2019.10772. Epub 2019 Oct 25. PMID 31661120
- [Background] Boland EG, Bennett MI, Allgar V, Boland JW. Cannabinoids for adult cancer-related pain: systematic review and meta-analysis. BMJ Support Palliat Care. 2020 Mar;10(1):14-24. doi: 10.1136/bmjspcare-2019-002032. Epub 2020 Jan 20. PMID 31959586
- [Background] Imanaka K, Tominaga Y, Etropolski M, Ohashi H, Hirose K, Matsumura T. Ready conversion of patients with well-controlled, moderate to severe, chronic malignant tumor-related pain on other opioids to tapentadol extended release. Clin Drug Investig. 2014 Jul;34(7):501-11. doi: 10.1007/s40261-014-0204-3. PMID 24906437
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Background] Freynhagen R, Baron R, Tolle T, Stemmler E, Gockel U, Stevens M, Maier C. Screening of neuropathic pain components in patients with chronic back pain associated with nerve root compression: a prospective observational pilot study (MIPORT). Curr Med Res Opin. 2006 Mar;22(3):529-37. doi: 10.1185/030079906X89874. PMID 16574036
- [Background] Lee SH, Min YS, Park HY, Jung TD. Health-related quality of life in breast cancer patients with lymphedema who survived more than one year after surgery. J Breast Cancer. 2012 Dec;15(4):449-53. doi: 10.4048/jbc.2012.15.4.449. Epub 2012 Dec 31. PMID 23346175
- [Background] Rehberg B, Mathivon S, Combescure C, Mercier Y, Savoldelli GL. Prediction of Acute Postoperative Pain Following Breast Cancer Surgery Using the Pain Sensitivity Questionnaire: A Cohort Study. Clin J Pain. 2017 Jan;33(1):57-66. doi: 10.1097/AJP.0000000000000380. PMID 27922844
- [Background] Handelsman L, Cochrane KJ, Aronson MJ, Ness R, Rubinstein KJ, Kanof PD. Two new rating scales for opiate withdrawal. Am J Drug Alcohol Abuse. 1987;13(3):293-308. doi: 10.3109/00952998709001515. PMID 3687892
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Pain: clinical manual for nursing practice Pain: clinical manual for nursing practice Margo McCaffery Alexander Beebe Mosby Yearbook UK pound17.25 0 7234 1992 2. Nurs Stand. 1994 Dec 7;9(11):55. doi: 10.7748/ns.9.11.55.s69. PMID 27527475
- See also: Note for Guidance on Clinical Safety Data Management: Definitions and Standards for Expedited Reporting (CPMP/ICH/377/95). Annotated with TGA comments,. 2001. — https://www.tga.gov.au/sites/default/files/ich37795.pdf
- See also: VA Evidence-based Synthesis Program Reports. In Benefits and Harms of Cannabis in Chronic Pain or Post-traumatic Stress Disorder: A Systematic Review, Department of Veterans Affairs (US): Washington (DC), 2017. — https://www.ncbi.nlm.nih.gov/books/NBK476449/